CLINICAL TRIAL: NCT03130075
Title: Reliability and Validity of the Turkish Version of Caregiver Functional Use Survey (CFUS)
Acronym: VERSION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ramazan Yildiz, research assisstant, Gazi University
Other Study IDs: E.150100
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Increasing the number of Turkish version of the questionnaire evaluating hand use, adding the scales that evaluate the selective movements of the upper limb to the evaluations will increase the variety of evaluation methods.

The purpose of this study is to evaluate the validity and reliability of the Turkish version of the Caregiver Functional Use Survey (CFUS)

DETAILED DESCRIPTION:
CFUS was designed to assess caregivers' perceptions of how much and how well their child used the involved upper extremity.

Children's upper extremity functions will be assessed with a Jebsen Taylor Hand Function Test. Their family will be asked to fill the CFUS.

Compare the relationship between Jebsen-Taylor Hand Function Test and Turkish Version CFUS. Investigate the internal consistency of Turkish-version of CFUS by using Cronbach's alpha coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 3-15 years
* Diagnosed as Cerebral Palsy (Hemiplegia)
* Literate in Turkish language and can complete the questionnaire by primer caregiver

Exclusion Criteria:

* Cannot understand the questionnaire by themselves.
* Participants had a botulinum toxin injection within the last 6 months
* Any surgical correction within the last year

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Hemiplegia Cerebral Palsy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-07-25 (Estimated); Study Completion 2017-08-25 (Estimated)

PRIMARY OUTCOMES:
Validity of Caregiver Functional Use Survey (CFUS) | 8 week
  Compare the relationship between Jebsen-Taylor Hand Function Test and Turkish Version CFUS

SECONDARY OUTCOMES:
Reliability of CFUS | 8 week
  Investigate the internal consistency of Turkish-version of CFUS by using Cronbach's alpha coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Elbasan, Study Chair — Study chair
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No